CLINICAL TRIAL: NCT04846868
Title: A Phase III Randomized, Double-blind, Placebo-controlled Parallel Group Trial to Examine the Efficacy and Safety of Iclepertin Once Daily Over 26 Week Treatment Period in Patients With Schizophrenia (CONNEX-1)
Brief Title: Clinical Trial of Iclepertin Effect on Cognition and Functional Capacity in Schizophrenia (CONNEX-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1346-0011; 2020-003760-11 (EudraCT Number)
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iclepertin 10 mg (Experimental): Patients with schizophrenia took orally once a day one 10 milligram (mg) tablet of iclepertin.
  Interventions: Drug: Iclepertin
- Placebo-matching Iclepertin 10 mg (Placebo Comparator): Patients with schizophrenia took orally once a day one tablet of placebo-matching iclepertin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iclepertin — One 10 milligram (mg) tablet once a day.
  Arms: Iclepertin 10 mg
Drug: Placebo — One tablet once a day.
  Arms: Placebo-matching Iclepertin 10 mg

SUMMARY:
This study is open to adults with schizophrenia. Schizophrenia can affect the way a person thinks, their memory and their mental functioning. Examples include struggling to remember things, or to read a book or pay attention to a movie. Some people have difficulty calculating the right change or planning a trip so that they arrive on time. The purpose of this study is to find out whether a medicine called Iclepertin improves learning and memory in people with schizophrenia.

Participants are put into two groups randomly, which means by chance. One group takes Iclepertin tablets and the other group takes placebo tablets. Placebo tablets look like Iclepertin tablets but do not contain any medicine. Participants take a tablet once a day for 26 weeks. In addition, all participants take their normal medication for schizophrenia.

During this time, doctors regularly test learning and memory of the participants by use of questionnaires, interviews, and computer tests. The results of the mental ability tests are compared between the groups.

Participants are in the study for about 8 months and visit the study site about 14 times. During this time, doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

1. Patients must be capable of providing signed and dated written informed consent by date of Visit 1 in accordance with ICH Harmonized Tripartite Guideline for Good Clinical Practice (ICH-GCP) and the local legislation prior to the admission to the trial.
2. Male or female patients who are 18-50 years (inclusive) of age at time of consent.
3. Diagnosis of schizophrenia utilizing Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) with the following clinical features:

   * Outpatient, clinically stable and in the residual (non-acute) phase of their illness.
   * No hospitalization or increase in level of psychiatric care due to worsening of schizophrenia within 12 weeks prior to randomization.
   * Positive and Negative Syndrome Scale (PANSS) score: items P1, P3-P6 ≤ 5 and item P2 and P7 ≤ 4 at Visit 1, and confirmed at Visit 2.
4. Patients should have functional impairment in day-to-day activities such as difficulties following conversation or expressing themselves, difficulties to stay focused, difficulties to remember instructions, what to say or how to get to places, per investigator judgement.
5. Patients maintained on current antipsychotic treatment (minimum 1 and maximum 2 antipsychotics, but clozapine is not allowed) for at least 12 weeks and on current dose for at least 35 days prior to randomization.

   -- For patients on two antipsychotics, at least one antipsychotic must be within the approved label dose range. The second antipsychotic must not exceed the maximum daily dose per local label.

   Note: If the total dose is stable, different dosage forms of the same antipsychotic treatment will be considered as one antipsychotic.
6. Patients with any other concomitant psychoactive medications (except for anticholinergics) need to be maintained on same drug for at least 12 weeks and on current dose/ regimen for at least 35 days prior to randomization.

   * Maximum daily benzodiazepine load of up to 1 mg lorazepam-equivalent.
   * For any other psychoactive medications, doses cannot exceed the maximum daily dose per local label.
7. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per Non-Clinical Safety Studies for the Conduct of Human Clinical Trials and Marketing Authorization for Pharmaceuticals (ICH M3 (R2)) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the protocol. Such methods should be used throughout the trial, and for a period of at least 35 days after last trial drug intake, and the patient must agree to periodic pregnancy testing during participation in the trial.
8. Have a study partner, defined as any person either private or professional who knows the patient well, has been capable of interacting with the patient on regular basis, and preferably consistent throughout the study.

   * The study partner must interact with the subject a minimum 1 hour per week and, preferably, at least 2 times a week. At least one interaction per week should be in person.
   * The study partner must have educational achievement of minimum 8th grade.
   * Professional study partners (e.g. study nurse, social worker etc.) are allowed if not involved in administration of any of the protocol assessments.

Further inclusion criteria apply.

Exclusion criteria

1. Participant with current DSM-5 diagnosis other than Schizophrenia, including but not limited to bipolar, schizoaffective, major depressive disorder etc. Mini International Neuropsychiatric Interview (M.I.N.I.) for Psychotic disorders should be used for guidance.
2. Cognitive impairment due to developmental, neurological (e.g., epilepsy, stroke) or other disorders including head trauma, or patients with dementia or epilepsy.
3. Severe movement disorders

   * Leading to cognitive impairment (e.g. Parkinson dementia), or
   * Interfering with the efficacy assessments, or
   * Due to antipsychotic treatment that cannot be controlled with low dose anticholinergic treatment (equal to maximum 1 mg benztropine twice daily).
4. Any suicidal behavior in the past 1-year prior to screening and during the screening period.
5. Suicidal ideation of type 5 in the Columbia Suicide Severity Rating Scale (C-SSRS) (i.e. active suicidal thought with plan and intent) in the past 3 months prior to screening and up to and including Visit 2.

   -- Patients with Suicidal Ideation type 4 in the C-SSRS (i.e. active suicidal thought with intent but without specific plan), within 3 months prior to screening and up to and including Visit 2, can be randomized in the study, if assessed and documented by a licensed mental health professional that there is no immediate risk of suicide.
6. History of moderate or severe substance use disorder (other than caffeine and nicotine), as defined in DSM-5 within the last 12 months prior to informed consent.
7. Positive urine drug screen at Visit 1 based on central lab test.
8. Patients who were treated with any of the following within 6 months prior to randomization:

   * Clozapine
   * Stimulants (e.g. methylphenidate, dextroamphetamine, modafinil)
   * Ketamine or esketamine
   * Electroconvulsive therapy (ECT) or Modified ECT Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 620 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (116):
- United States (18):
  - Collaborative Neuroscience Network, LLC (CNS), Garden Grove, California
  - Omega Clinical Trials,LLC, La Habra, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Velocity Clinical Research-Santa Ana-68902, Santa Ana, California
  - Institute of Living, Hartford, Connecticut
  - San Marcus Research Clinic, Inc., Miami, Florida
  - CCM Clinical Research Group, LLC-Miami-68482, Miami, Florida
  - Atlanta Center, Atlanta, Georgia
  - University at Buffalo, The State University of New York, Buffalo, New York
  - Richmond Behavioral Associates-Staten Island-68636, Staten Island, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - PeaceHealth Medical Group, Eugene, Oregon
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Houston Mind and Brain, Houston, Texas
  - Core Clinical Research, Everett, Washington
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia
- Brazil (7):
  - CPN - Centro de Estudos em Neurociências, Belo Horizonte
  - Hospital das Clinicas da Universidade Federal de Minas Gerais (HCUFMG), Belo Horizonte,Minas Gerais
  - Hospital Sao Jose, Criciúma
  - Trial Tech- Tecnologia em pesquisa com medicamentos, Curitiba
  - J A Serviços Médicos Ltda/ Instituto Goiano de Neuropisquiatria, Goiânia
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
  - BR Trials, São Paulo
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - OCT Research ULC, Kelowna, British Columbia
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
- China (13):
  - The sixth People's Hospital of Hebei Province, Baoding
  - Peking University Sixth Hospital, Beijing
  - Beijing HuiLongGuan Hospital, Beijing
  - The Second People's Hospital of Hunan Province (Brain Hospital of Hunan Province), Changsha
  - The Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Shandong Daizhuang Hospital, Jining
  - The First Affilliated Hospital Of Kunming of Medical College, Kunming
  - The Affilicated Kangning Hospital of Ningbo University, Ningbo
  - Shanghai Mental Health Center, Shanghai
  - Tongji Hospital, Tongji University, Shanghai
  - Wuxi mental health center, Wuxi
  - The Second Affiliated Hospital of Xinxiang Medical Univ., Xinxiang
- Colombia (5):
  - Centro de Investigación y Proyectos en neurociencia CIPNA, Barranquilla
  - E.S.E Hospital Mental de Antioquia, Bello
  - Instituto Colombiano del Sistema Nervioso- Clínica Montserrat, Bogotá
  - Centro de Investigaciones del Sistema Nervioso SAS- Grupo Cisne SAS, Bogotá
  - Psynapsis Salud Mental S.A., Pereira
- Germany (4):
  - Zentrum für klinische Forschung Dr. med. I. Schöll GmbH, Bad Homburg
  - Praxis Dr. Hahn, Berlin, Berlin
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Neurologie und Psychiatrie / Psychotherapie, Westerstede
- Greece (7):
  - Eginition Hospital, Athens
  - "Attikon" University General Hospital of Attica, Chaïdári
  - Psychiatric Hospital of Attica, Haidari
  - AX Mental Health Clinic, Heraklion
  - General Oncology Hospital "Agioi Anargyri", Nea Kifissia
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Italy (5):
  - ASST degli Spedali Civili di Brescia, Brescia
  - A.O. Fatebenefratelli, Milan
  - Ist. San Raffaele Turro, Milan
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano (TO)
  - A.O.U. Senese, Siena
- Japan (30):
  - Hotei Hospital, Aichi, Konan
  - Japan Institute for Health Security National Kohnodai Medical Center, Chiba, Ichikawa
  - Mental Clinic Sakurazaka, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kuramitsu Hospital, Fukuoka, Fukuoka
  - Shiranui Hospital, Fukuoka, Omuta
  - Obihiro-Kosei General Hospital, Hokkaido, Obihiro
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - St. Marianna University Hospital, Kanagawa, Kawasaki
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Yokohama Onoecho Clinic, Kanagawa, Yokohama
  - Hino Hospital, Kanagawa, Yokohama
  - Kochi Health Sciences Center, Kochi, Kochi
  - National Hospital Organization Maizuru Medical Center, Kyoto, Maizuru
  - Tohoku University Hospital, Miyagi, Sendai
  - Shounan Hospital, Nagano, Matsumoto
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - National Hospital Organization Hizen Psychiatric Medical Center, Saga, Kanzaki-gun
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Nishi Kumagaya Hospital, Saitama, Kumagaya
  - Sho Midori Hospital, Saitama, Saitama
  - Dokkyo Medical University Hospital, Tochigi, Shimotsuga-gun
  - Tokushima University Hospital, Tokushima, Tokushima
  - National Center of Neurology and Psychiatry, Tokyo, Kodaira
  - Asuka Hospital, Tokyo, Machida
  - Showa University Karasuyama Hospital, Tokyo, Setagaya
  - Shinjuku East Mental Clinic, Tokyo, Shinjuku-ku
  - Ohwa Mental Clinic, Tokyo, Toshima-ku
  - Yamaguchi University Hospital, Yamaguchi, Ube
  - University of Yamanashi Hospital, Yamanashi, Chuo
- Mexico (6):
  - Clinica Cemelli, Guadalajara
  - GabiPros S.C., Mexico City
  - Instituto Nacional de Neurologia y Neurocirugia, Mexico City
  - Medical Care & Research SA de CV, Mérida
  - CIT-Neuropsique S.C, Monterrey
  - Instituto de Informacion e Investigacion en Salud Mental A.C. (INFOSAME)., Monterrey
- North Shore Hospital, Takpuna Auckland, New Zealand
- Norway (2):
  - Sykehuset Østfold HF, avd. Moss, Moss
  - Akershus Universitetssykehus HF, Oslo
- Philippines (2):
  - St. Paul's Hospital-Iloilo City-40765, Iloilo City
  - Philippine General Hospital, Manila, Philippines
- Poland (5):
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - Central Teaching Hospital of the Medical University of Lodz, Lodz
  - Individual Specialist Medical Practice Filip Rybakowski, Poznan
  - Institute of Psychiatry and Neurology in Warsaw, Warsaw
  - Clinhouse, Zabrze
- Sweden (2):
  - Psykiatriska Kliniken, Helsingborg
  - Akademiska sjukhuset, Uppsala
- Turkey (Türkiye) (5):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara University Medical School, Ankara
  - Istanbul University, Istanbul
  - Dokuz Eylul Universitesi Psikiyatri A.B.D., Izmir
  - Celal Bayar Universitesi Tip Fakultesi, Manisa

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Keefe RSE, Harvey PD, Correll CU, Falkai P, Hashimoto N, Klein H, Krystal JH, Marder S, Medalia A, Sumiyoshi T, Wang G, Zhang H, Blahova Z, Bichard-Sall I, English BA, Fu E, Gruenenfelder F, Groeschl M, Kimura K, Tang W, von der Goltz C, Fowler C. Efficacy and safety of iclepertin for cognitive impairment associated with schizophrenia (CONNEX programme): results from three phase 3 randomised controlled trials. Lancet Psychiatry. 2025 Dec;12(12):906-920. doi: 10.1016/S2215-0366(25)00296-2. PMID 41233083
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, placebo-controlled, double-blind, multicenter, multinational, 26-week, parallel group trial. Patients could roll-over to safety follow-up extension trial (study 1346-0014). A dedicated ocular sub-study was implemented in several countries participating in the trial to investigate the ocular safety of iclepertin in patients with schizophrenia.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Started | 312 | 308
Treated | 312 | 307
Ocular safety sub-study | 26 | 22
Completed | 266 | 273
Not Completed | 46 | 35
Not completed — Adverse Event | 12 | 11
Not completed — Protocol deviation | 6 | 2
Not completed — Perceived lack of efficacy | 3 | 2
Not completed — Change of residence | 2 | 3
Not completed — Burden of study procedures | 1 | 1
Not completed — No reason available | 2 | 5
Not completed — Other reason listed | 20 | 10
Not completed — Not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set: all patients randomized into the trial, regardless of whether a patient was treated with trial medication. One patient was randomized in error and discontinued from the trial before the start of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg | Total
Number analyzed (Participants) | 312 | 307 | 619
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (9.0) | 33.8 (8.8) | 34.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 104 | 211
  Male | 205 | 203 | 408
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 123 | 123 | 246
  Not Hispanic or Latino | 189 | 184 | 373
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 53 | 63 | 116
  Asian | 88 | 97 | 185
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 21 | 19 | 40
  White | 139 | 122 | 261
  More than one race | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
MATRICS Consensus Cognitive Battery (MCCB) overall composite T-score [Mean (Standard Deviation); unit: Units on a scale] — MCCB comprises 10 tests, which assess 7 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The larger the MCCB overall composite T-score, the better patient cognition. A mean T-score of 50 and a standard deviation of 10 reflects the T-score on a general population.
  Units on a scale | 28.6 (13.7) | 28.8 (14.0) | 28.7 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Composite T-score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) After 26 Weeks of Treatment
Description: MCCB comprises 10 tests, which assess 7 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The larger the MCCB overall composite T-score, the better patient cognition. A mean T-score of 50 and a standard deviation of 10 reflects the general population.
  The estimated treatment effect included the effect of any concomitant therapies for all randomized patients on on-treatment periods. On-treatment is defined as the period of first drug administration/first resumed dose after interruption until last drug administration + REP (residual effect period).
  The change from baseline was analyzed with a MMRM (mixed-effects model for repeated measures) with the fixed effects: treatment at each visit, stratification factor using the screening MCCB overall composite T-score, and baseline MCCB overall composite T-score at each visit. Visit was the repeated measure.
Time Frame: MMRM included measurements at baseline, Week 12, and Week 26. Change from baseline values at Week 26 is reported.
Population: Randomized set: all patients randomized into the trial, regardless of whether a patient was treated with trial medication. Patients on an off-treatment period due to temporary treatment discontinuation or early permanent treatment discontinuation were excluded from the analysis according to the strategy to handle intercurrent events defined in the statistical analysis plan. One patient was randomized in error and discontinued from the trial before the start of trial medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Number analyzed (Participants) | 288 | 294
Units on a scale | 2.283 (0.3094) | 2.22 (0.3065)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo-matching Iclepertin 10 mg; MMRM, including the fixed effects: treatment at each visit, stratification factor using the screening MCCB overall composite T-score, and baseline MCCB overall composite T-score at each visit. Visit was the repeated measure with an unstructured covariance structure to model the within-patient measurements; Test type: Superiority — The estimated treatment effect included the effect of any concomitant therapies for all randomized patients on on-treatment periods; p = 0.8854, Mixed Models Analysis — Null hypothesis: The adjusted mean change from baseline to Week 26 in MCCB overall composite T-score in iclepertin 10mg is worse than or equal to that in placebo. one-sided p< 0.025 required for testing subsequent key secondary endpoint hypotheses; Mean Difference (Net) = 0.063, 95% CI 2-sided [-0.793 to 0.918], Standard Error of Mean 0.4355 — Iclepertin 10 mg versus Placebo

2. Secondary Outcome: Key Secondary Endpoint: Change From Baseline in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Total Score After 26 Weeks of Treatment
Description: The SCoRS is an interview based- assessment tool to evaluate the cognitive function of individuals with schizophrenia that incorporates the input of the patient, the caregiver and the interviewer. It is composed of 20 items on a 7-point Likert scale, ranging from 20 to 140 points, where a higher score indicates a greater cognitive impairment.
  The estimated treatment effect included the effect of any concomitant therapies and partner change in SCoR assessment for all randomized patients on-treatment. On-treatment is defined as the period of 1st drug administration/1st resumed dose after interruption until last drug administration + REP.
  The change from baseline was analyzed with mixed-effects model for repeated measures (MMRM) with the fixed effects: treatment at each visit, stratification factor using the screening MCCB overall composite T-score, and baseline MCCB overall composite T-score at each visit. Visit was treated as the repeated measure.
Time Frame: MMRM included measurements at baseline, Week 12, and Week 26. Change from baseline values at Week 26 is reported.
Population: Randomized set: all patients randomized into the trial, regardless of whether a patient was treated with trial medication. Patients on an off-treatment period due to temporary treatment discontinuation or early permanent treatment discontinuation were excluded from the analysis of this endpoint according to the strategy to handle intercurrent events defined in the statistical analysis plan. One patient was randomized in error and discontinued from the trial before the start of trial medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Number analyzed (Participants) | 292 | 292
Units on a scale | -5.246 (0.4150) | -5.480 (0.4140)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo-matching Iclepertin 10 mg; MMRM including the fixed effects: treatment at each visit, stratification factor using the screening MCCB overall composite T-score, and baseline MCCB overall composite T-score at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements; Test type: Other — The estimated treatment effect included the effect of any concomitant therapies and partner change in SCoR assessment for all randomized patients on-treatment; p = 0.6902, Mixed Models Analysis; Mean Difference (Net) = 0.234, 95% CI 2-sided [-0.918 to 1.386], Standard Error of Mean 0.5867 — Iclepertin 10 mg versus Placebo

3. Secondary Outcome: Key Secondary Endpoint: Change From Baseline to Week 26 in the Adjusted Total Time T-score in the Virtual Reality Functional Capacity Assessment Tool (VRFCAT)
Description: The VRFCAT is a computerized assessment measuring the functional capacity of an individual to perform everyday tasks. It generates a composite score based on the amount of time taken to complete the tasks. The lower the VRFCAT T-score, the better patient's functional capacity. A mean T-score of 50 and a standard deviation of 10 reflects the T-score in a general population.
  The estimated treatment effect included the effect of any concomitant therapies for all randomized patients on-treatment. On-treatment is defined as the period of 1st drug administration/1st resumed dose after interruption until last drug administration + REP.
  The change from baseline was analyzed with MMRM with the fixed effects: treatment at each visit, stratification factor using the screening MCCB overall composite T-score, and baseline MCCB overall composite T-score at each visit. Visit was treated as the repeated measure.
Time Frame: MMRM included measurements at baseline, Week 12, and Week 26. Change from baseline values at Week 26 is reported.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Number analyzed (Participants) | 292 | 296
Units on a scale | 3.108 (0.8089) | 3.652 (0.8018)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo-matching Iclepertin 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other — The estimated treatment effect included the effect of any concomitant therapies for all randomized patients on-treatment; p = 0.6334, Mixed Models Analysis; Mean Difference (Net) = -0.543, 95% CI 2-sided [-2.780 to 1.694], Standard Error of Mean 1.1388 — Iclepertin 10 mg vs. placebo

4. Secondary Outcome: Change From Screening Visit 1a in Patient Reported Experience of Cognitive Impairment in Schizophrenia (PRECIS) Total Score at Week 24
Description: The Patient Reported Experience of Cognitive Impairment in Schizophrenia (PRECIS) score evaluates how cognitive difficulties impact the daily life of individuals with schizophrenia. It is composed of 28 items on a 5-category Likert scale (1=not at all/not at all hard, 5=very much/very hard), and the total score was derived by calculating the average score of the first 26 items, where higher scores mean a worse patient experience.
  The estimated treatment effect included the effect of any concomitant therapies for all randomized patients on-treatment. On-treatment is defined as the period of 1st drug administration/1st resumed dose after interruption until last drug administration + REP.
  The change from baseline was analyzed with MMRM with the fixed effects: treatment at each visit, stratification factor using the screening MCCB overall composite T-score, and baseline MCCB overall composite T-score at each visit. Visit was treated as the repeated measure.
Time Frame: MMRM included measurements at Visit 1a (Week -2/Week -1), Week 15, and Week 24. Change from Visit 1a values at Week 24 is reported.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Number analyzed (Participants) | 291 | 292
Units on a scale | -0.258 (0.0317) | -0.305 (0.0316)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo-matching Iclepertin 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.2902, Mixed Models Analysis; Mean Difference (Net) = 0.047, 95% CI [-0.041 to 0.135], Standard Error of Mean 0.0448 — Iclepertin 10 mg vs Placebo

5. Secondary Outcome: Change From Baseline in the T-score of the Number of Correct Responses on Tower of London at Week 26
Description: The Tower of London (ToL) evaluates executive functioning, reasoning, problem-solving, and goal-directed behavior. It measures the number of correct responses in solving an exercise that consists on moving colored balls to match a target configuration. The higher the ToL T-score, the better patient's cognitive function. A mean T-score of 50 and a standard deviation of 10 reflects the T-score in a general population.
  The estimated treatment effect included the effect of any concomitant therapies for all randomized patients on-treatment. On-treatment is defined as the period of 1st drug administration/1st resumed dose after interruption until last drug administration + REP.
  The change from baseline comparing the groups was analyzed using analysis of covariance (ANCOVA) model including treatment, stratification factor of screening MCCB overall composite T-score, and baseline number of correct responses on Tower of London T-score.
Time Frame: At baseline and at Week 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Number analyzed (Participants) | 273 | 279
Units on a scale | 1.103 (0.6547) | 0.475 (0.6477)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo-matching Iclepertin 10 mg; ANCOVA model including treatment, stratification factor of screening MCCB overall composite T-score, and baseline number of correct responses on Tower of London T-score; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.4956, ANCOVA; Mean Difference (Net) = 0.628, 95% CI 2-sided [-1.181 to 2.437] — Iclepertin 10 mg vs. Placebo

6. Secondary Outcome: Ocular Safety Sub-study: Humphrey Visual Field 24-2 Swedish Interactive Thresholding Algorithm (SITA) Standard
Description: The Humphrey Visual Field 24-2 SITA Standard is a diagnostic test to measure visual fields, or perimetry. The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a central spot. The perception of these lights is charted and then compared to results of a healthy eye at the same age of the patient to determine if any damage has occurred. The tests ranks from 0 to 100%, where 0 means no vision and 100 means perfect vision.
Time Frame: At baseline and at Week 24.
Population: Ocular sub-study set: all treated patients who consented to participate in the ocular sub-study. Only patients with measurements were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Number analyzed (Participants) | 23 | 21
Units on a scale
  Left eye - baseline | 93.83 (8.82) | 95.62 (5.56)
  Right eye - baseline | 95.87 (5.60) | 95.87 (5.60)
  Left eye - Week 24 | 94.48 (10.69) | 96.00 (6.58)
  Right eye - Week 24 | 95.83 (5.69) | 95.83 (5.69)

7. Secondary Outcome: Ocular Safety Sub-study: Central Retinal Thickness as Measured by Spectral Domain Optical Coherence Tomography (SD-OCT)
Description: The central retinal thickness for both eyes was measured by high-definition optical coherence tomography (spectral domain OCT), which evaluates the retinal and sub-retinal structures of both eyes.
Time Frame: At baseline and at Week 24.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
Number analyzed (Participants) | 25 | 21
micrometer
  Left eye - baseline | 231.52 (26.51) | 230.38 (26.64)
  Right eye - baseline | 233.12 (31.03) | 235.00 (25.45)
  Left eye - Week 24: number analyzed (Participants) | 24 | 19
  Left eye - Week 24 | 237.67 (27.32) | 236.10 (25.96)
  Right eye - Week 24: number analyzed (Participants) | 23 | 19
  Right eye - Week 24 | 235.46 (27.81) | 240.49 (26.89)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization until individual end of study. Up to 246 days. Adverse event reporting: From first drug administration to last drug administration, plus residual effect period OR from first drug administration until first drug administration on the extension trial 1346-0014. Up to 230 days.
Description: Treated Set (TS): all patients who signed informed consent and were treated with at least one dose of the trial medication.
Arm/Group | Iclepertin 10 mg | Placebo-matching Iclepertin 10 mg
All-Cause Mortality (participants affected / at risk) | 1/312 | 1/307
Serious Adverse Events (participants affected / at risk) | 12/312 | 16/307
Other Adverse Events (participants affected / at risk) | 81/312 | 91/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iclepertin 10 mg (N=312) | Placebo-matching Iclepertin 10 mg (N=307)
Myocardial infarction (Cardiac disorders) | 0 | 1
Central serous chorioretinopathy (Eye disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 5 | 6
Suicidal ideation (Psychiatric disorders) | 2 | 6
Suicide attempt (Psychiatric disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iclepertin 10 mg (N=312) | Placebo-matching Iclepertin 10 mg (N=307)
Influenza (Infections and infestations) | 8 | 16
Nasopharyngitis (Infections and infestations) | 21 | 16
Upper respiratory tract infection (Infections and infestations) | 16 | 11
Headache (Nervous system disorders) | 22 | 27
Insomnia (Psychiatric disorders) | 10 | 16
Schizophrenia (Psychiatric disorders) | 17 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT04846868/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT04846868/SAP_001.pdf